CLINICAL TRIAL: NCT05583487
Title: Multidisciplinary Teamwork Perceptions When Mobilizing Ventilated Neurosurgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Adrianna Lall, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: STU-2022-0903
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Multidisciplinary Communication
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study will consist of a quasi-experimental research design to examine causality between two or more variables by comparing groups following an intervention. Although the intervention itself will be randomly assigned/administered to each of the multidisciplinary groups for this proposed research study, true randomization of participants cannot be achieved. This is primarily due to each patient having a pre-assigned multidisciplinary care team for each shift. Changing this patient assignment would compromise patient safety while interfering with continuity of care and workflow, which hospital units strive to achieve. By applying the purpose and elements of a quasi-experimental approach to this proposed research study, researchers can determine if an intervention/active independent variable consisting of a nurse-led mobility protocol, has an effect on the outcome measure of teamwork perceptions , which will serve as dependent variables.
Who Masked: Care Provider
Masking Description: All teams will be asked to progressively mobilize the ventilated neurosurgery patient they are assigned to during the shift. Each team will be blinded to whether or not they will be utilizing the nurse-led mobility protocol or standard mobility procedures until arrival at the patient's room during the assigned mobility time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/non-experimental group (Active Comparator): The control/nonexperimental group will consist of multidisciplinary teams, who will not be given the nurse-led protocol and will be asked to mobilize the assigned ventilated neurosurgery patient according the facility's standard mobility procedures.
  Interventions: Other: Standard of Care
- Experimental/interventional group (Experimental): The experimental/interventional group will consist of multidisciplinary teams who will use a given nurse-led protocol (intervention) to mobilize the assigned patient.
  Interventions: Other: Nurse-led progressive mobility protocol

INTERVENTIONS:
Other: Nurse-led progressive mobility protocol — The nurse-led mobility progression protocol incorporates a checklist for four primary team members belonging to each discipline to follow before, during, and after providing mobility for each patient. It outlines steps to progress patient mobility from in-bed mobility activities to out-of-bed activities as tolerated. This protocol intervention was created and designed based upon a review of previously conducted studies' interventions and findings, as well as expert guidelines established in the literature. Furthermore, multidisciplinary experts at the medical center who work with ventilated neurosurgery patients were consulted to form the protocol to further establish hemodynamic, neurological, respiratory, and physiological patient safety parameters. This intervention has not been implemented in previous studies and will be piloted for this study.
  Other Names: nurse-led protocol
  Arms: Experimental/interventional group
Other: Standard of Care — For the purposes of the current study, the control group of multidisciplinary teams requested to mobilize the ventilated neurosurgery patient, may also consist of the primary nurse, RT, PT, and PCT. They will be asked to progressively mobilize the patient to the best of their ability according to standard of care procedures, incorporating any resources the medical center provides including, but not limited to, written information, equipment, ThinkLift, etc.
  Arms: Control/non-experimental group

SUMMARY:
The purpose of this research study is to decide if using a nurse-led mobility protocol affects teamwork perceptions, when mobilizing ventilated neurosurgery patients. Participants will mobilize ventilated neurosurgery patients according to either facility standard procedures or a piloted nurse-led mobility protocol. Each selected patient will be mobilized once during his/her hospitalization for the purposes of this study. Patient mobility may take up to 1 hour. Following this, participating staff will be asked to complete a survey used to measure teamwork perceptions. Participants will be given up to 30 minutes to complete the survey. Total study duration is 3 months.

ELIGIBILITY:
Inclusion Criteria:

* adult (18 years of age or older)
* male or female registered nurses or licensed vocational nurses, patient care technicians, respiratory therapists, and physical therapists
* currently employed by the medical center
* currently care for neurosurgery patients in a part time or full-time capacity
* may work during day shift and/or night shift hours.

Exclusion Criteria:

* staff members employed by an agency outside of the medical center
* staff not routinely assigned to care for neurosurgery patients on the neurosurgical ICU (float pool staff)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Teamwork perceptions | Will take each participant no more than 30 minutes to complete. Each participant will take this once following each patient mobility instance.
  Will be measured using the reliable and valid Nursing Teamwork Survey (NTS) established by Beatrice Kalisch, PhD. The NTS is composed of items with Likert-type scale ranging from 1-5. Higher scores indicate more positive perceptions of teamwork, while lower scores indicate more negative perceptions of teamwork. This scale has been tested and has good psychometric properties including adequate validity and reliability. The minimum total score is 33, while the highest possible score is 165 per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Adrianna Lall, Principal Investigator — University of Texas at Arlington
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No